CLINICAL TRIAL: NCT01703338
Title: Clinical and Biomechanics Research in Core Muscles After Lumbar Fusion Surgery
Status: Terminated | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112117RIC
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Lumbar Fusion; Lumbar Spinal Fusion Surgery
Keywords: assessment model; biomechanical changes; functional activities; magnetic resonance imaging (MRI); causal relationship; core muscles activation pattern; pathological changes; early rehabilitation; core stability exercise; minimally invasive lumbar spinal fusion surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar spinal surgery: The study included participants who were diagnosed by a neurological surgeon and received lumbar surgery according to relevant imaging findings

SUMMARY:
Lumbar fusion has been widely used for spinal disorders when conservative treatment has failed. However, a number of studies have reported that the rate of re-operation is high for lumbar fusion surgery. Swelling, atrophy or fat infiltration of the paraspinal muscles at the surgery site can cause weakness and pain. After fusion, the range of motion is constrained at the fused spine and might facilitate compensative movement of the adjacent levels and increase degeneration rate of the spine.

Evidence has shown that core muscles play an important role to stabilize and support the spine. Whether core stability exercise can enhance spinal stability after lumbar fusion surgery remains unclear. Therefore, the overall goal of this proposed research is to investigate how core muscles affect outcomes after lumbar spinal fusion. The investigators will explore this issue hierarchically and systematically in 3-year duration.

ELIGIBILITY:
Inclusion Criteria:

1. ages between 20 and 85 years,
2. back pain and/or sciatica exceeding 12 weeks for which conservative treatment had failed to improve,
3. a primary diagnosis of spinal stenosis, spondylosis, degenerative or isthmic spondylolisthesis or degenerative disc disease, and
4. the patient selected for lumbar surgery

Exclusion Criteria:

1. mechanical back pain due to posture changes and cannot maintain an upright posture over 30 minutes;
2. segmental instability that includes isthmic spondylolisthesis, degenerative spondylolisthesis over 0.4 cm;
3. intervertebral angle reversal on dynamic radiographs; and
4. previous lumbar fusion, rheumatoid arthritis, and ankylosing spondylitis.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be recruited from the National Taiwan University Hospital and Far Eastern Memorial Hospital. The study is approved by the Institutional Medical Research Ethics Committees in both National Taiwan University Hospital and Far Eastern Memorial Hospital. Our neurological surgeon will response for subject screening and medical diagnose. According to the power analysis, fifty subjects will be enrolled in this study. The eligible subject will be given the subjects informed consent and sign it before the enrollment.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2018-12-24 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan